CLINICAL TRIAL: NCT01920178
Title: A Placebo Controlled, Randomized, Prospective Study to Evaluate the Efficacy and Safety of PinPointe FootLaser in Patients Who Have Failed Oral Terbinafine Treatment for Onychomycosis
Brief Title: Evaluation Study for the Efficacy and Safety of PinPointe FootLaser in Treatment for Onychomycosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial support of the Study withdrawn by Nuvolase, Inc ( PinPointe FootLaser) due to delayed start of the Study and inadequate subjects enrolled
Sponsor: Cambridge Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0860/08/11
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2016-07

CONDITIONS: Onychomycosis of Toenails

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PinPointe Foot Laser (Active Comparator): Active laser
  Interventions: Device: PinPointe Foot Laser
- Sham laser group (Sham Comparator): Treatment with only localizing (aiming) beam of Pinpointe Foot Laser
  Interventions: Device: PinPointe Foot Laser

INTERVENTIONS:
Device: PinPointe Foot Laser — Active Laser Treatment Group will receive active Pinpointe Foot Laser beam. Control Placebo Sham Laser Group will receive only the localizing (aiming) non-active beam of the Pinpointe Foot Laser

SUMMARY:
The purpose of this study is to assess the clinical efficacy and safety of the PinPointe Foot Laser device for the treatment of patients with onychomycosis who have been previously treated with oral Terbinafine and failed.

DETAILED DESCRIPTION:
This protocol is designed to demonstrate that the PinPointe FootLaser treatment is able to produce clinical improvement treating onychomycosis in patients who have previously taken Terbinafine and failed treatment. The duration of enrollment for each subject will be 2 years, with the expectation that this is the time period that will yield 100% reduction in the area of involved nail. Enrollment is competitive and we expect to enroll 40 patients at CHA.

The medical device that is the subject of this clinical trial is the PinPointe FootLaser, manufactured by NuvoLase, Inc. It is a pulsed Nd:Yag laser device that uses a proprietary pulse train, operating at 1064nm wavelength, with 100 μsec pulses. It received pre-market Section 510(k) clearance by the FDA and subsequent clearance for the treatment of onychomycosis in 2010.

Onychomycosis (OM), a fungal infection of the toes, is a major health problem around the world. It is estimated that there are more than 40 million sufferers with this condition in the USA. A recent European study showed that the prevalence of onychomycosis may be as high as 26.9%. Importantly, it is a particular problem that disproportionately affects diabetics. The main causative agent varies according to climate. Dermatophyte infections are common worldwide.

Preliminary in vitro and in vivo work has demonstrated the proof of principle that the PinPointe FootLaser device can kill microorganisms, including dermatophytes and other fungi, which infect the toenail. Based on these preliminary results, this study has been designed to demonstrate the efficacy and safety of the PinPointe FootLaser for clearing toenails, including those with onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* Previous treatment with at least 90 days of oral Terbinafine and completed the treatment at least 1 year ago
* Able to feel a Semmes-Weinstein monofilament at the tip of each toe
* Must have at least 50% involvement in at least one great toenail
* Must be willing and able to present for one treatment visit and two follow-up visits at 6 months and 12 months following initial treatment to photograph the nails
* Must be willing to apply topical antifungal to the skin surrounding the toes on a daily basis and be willing to spray shoes with an aerosolized antifungal on a weekly basis
* Must have dystrophic toenails which clinically appear to be mycotic
* Age ≥ 18 years and ≤ 70 years
* Willing to comply with study requirements, including regular nail debridement as indicated by the investigator
* Willing to provide informed consent to participate

Exclusion Criteria:

* Evidence of gangrene or non-palpable dorsalis pedis and posterior tibial pulses
* Capillary refill time greater than 5 seconds
* Patients who are severely immunocompromised (such as in AIDS, renal transplant regimens, immunosuppressed states consequent to malignancy or agents used in rendering oncologic care, or who suffer from end stage renal disease)
* Patients with documented diagnosis of psoriasis or lichen planus
* Actively treating fungal nails with a topical agent during the last 90 days prior to enrollment, including tea tree oil, antifungal nail polish, Penlac, fungoid tincture, or similar over-the-counter antifungal treatments
* Inability to follow treatment regimen or comply with follow-up schedules
* History of malignant melanoma or any forms of skin cancers
* Evidence of acute bacterial infections with or without cellulitis and/or purulence
* Treatment for onychocryptosis during the last 30 days or a history of recurrent onychocryptosis of at least 3 episodes in the last 12 months in which medical care such as resection by a podiatrist/physician, or use of antibiotics was rendered
* Toenail deformity associated with trauma, psoriasis or lichen planus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Heffernan, D.P.M., Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arrese JE, Pierard GE. Treatment failures and relapses in onychomycosis: a stubborn clinical problem. Dermatology. 2003;207(3):255-60. doi: 10.1159/000073086. PMID 14571066
- [Background] Elewski BE, Scher RK, Aly R, Daniel R 3rd, Jones HE, Odom RB, Zaias N, Jacko ML. Double-blind, randomized comparison of itraconazole capsules vs. placebo in the treatment of toenail onychomycosis. Cutis. 1997 Apr;59(4):217-20. PMID 9104548
- [Background] Gupta AK, Fleckman P, Baran R. Ciclopirox nail lacquer topical solution 8% in the treatment of toenail onychomycosis. J Am Acad Dermatol. 2000 Oct;43(4 Suppl):S70-80. doi: 10.1067/mjd.2000.109071. PMID 11051136
- [Background] Haneke E, Abeck D, Ring J. Safety and efficacy of intermittent therapy with itraconazole in finger- and toenail onychomycosis: a multicentre trial. Mycoses. 1998 Dec;41(11-12):521-7. doi: 10.1111/j.1439-0507.1998.tb00716.x. PMID 9919897
- [Background] Pollak R, Billstein SA. Efficacy of terbinafine for toenail onychomycosis. A multicenter trial of various treatment durations. J Am Podiatr Med Assoc. 2001 Mar;91(3):127-31. doi: 10.7547/87507315-91-3-127. PMID 11266494
- [Background] Potter LP, Mathias SD, Raut M, Kianifard F, Landsman A, Tavakkol A. The impact of aggressive debridement used as an adjunct therapy with terbinafine on perceptions of patients undergoing treatment for toenail onychomycosis. J Dermatolog Treat. 2007;18(1):46-52. doi: 10.1080/09546630600965004. PMID 17373090
- [Background] Scher RK, Tavakkol A, Sigurgeirsson B, Hay RJ, Joseph WS, Tosti A, Fleckman P, Ghannoum M, Armstrong DG, Markinson BC, Elewski BE. Onychomycosis: diagnosis and definition of cure. J Am Acad Dermatol. 2007 Jun;56(6):939-44. doi: 10.1016/j.jaad.2006.12.019. Epub 2007 Feb 16. PMID 17307276

RESULTS

PARTICIPANT FLOW:
Groups:
- PinPointe Foot Laser: Active laser
  PinPointe Foot Laser: Active Laser Treatment Group will receive active Pinpointe Foot Laser beam.
  Control Placebo Sham Laser Group will receive only the localizing (aiming) non-active beam of the Pinpointe Foot Laser
- Sham Laser Group: Treatment with only localizing (aiming) beam of Pinpointe Foot Laser
  PinPointe Foot Laser: Active Laser Treatment Group will receive active Pinpointe Foot Laser beam.
  Control Placebo Sham Laser Group will receive only the localizing (aiming) non-active beam of the Pinpointe Foot Laser
Period: Overall Study
Arm/Group | PinPointe Foot Laser | Sham Laser Group
Started | 5 | 2
Completed | 3 | 1
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PinPointe Foot Laser | Sham Laser Group | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.2) | 47.0 (2.8) | 44.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Measure Improvement in Target Toenails During the Study Period by Deeming a Clinical Success if Patient Experiences at Least a 50% Reduction in the Area of Involved Nail, Judged by the Clinician, and Judged by an Independent Evaluator.
Time Frame: 12 months
Population: Original grooved markings scored into the Target nails (hallux nails) on initial laser treatment visit to indicate most proximal aspect of fungal infection was intended to track the growth of the nail and to evaluate for improvement. Grooved markings did not survive after initial visit making it impossible to obtain valid primary endpoint data.
Arm/Group | PinPointe Foot Laser | Sham Laser Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Measure Clinical Improvement as Judged by the Patient and Determine Presence of Onychomycosis by PCR Analysis of Nail Samples
Time Frame: 12 months
Population: PCR lab analysis of nail samples obtained for each subject was not performed with the original study sponsor Nuvolase, Inc/ PinPointe withdrawing support for such analysis during the study.
Arm/Group | PinPointe Foot Laser | Sham Laser Group
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Number of Participants With Adverse Events During and Following Each Study Treatment
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | PinPointe Foot Laser | Sham Laser Group
Number analyzed (Participants) | 5 | 2
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events assessed both during and following each study treatment for all 10 toes with 2 laser passes over each clinically infected nail and one laser pass over each nail with no clinical signs of onychomycosis performed at each treatment.
Arm/Group | PinPointe Foot Laser | Sham Laser Group
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2

LIMITATIONS AND CAVEATS:
Withdrawal of financial support by Nuvolase, Inc in June, 2014 with very small enrollment of only 7 subjects ( 40 originally anticipated) led to loss of vital Primary and Secondary Outcome Measures with no reliable or interpretable data produced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes